CLINICAL TRIAL: NCT02671578
Title: Bispectral Index and Clinical Parameters Evaluation in Different Dental Procedures With Nitrous Oxide and Oxygen Sedation
Brief Title: Bispectral Index and Clinical Parameters Evaluation in Dental Procedures
Acronym: BIS-01
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Francisco Groppo (Other)
Collaborators: Faculty Sao Leopoldo Mandic Campinas (Other); pontifical catholic university - Rio de Janeiro (Unknown)
Responsible Party: Sponsor-Investigator, Francisco Groppo, Professor, University of Campinas, Brazil
Organization: University of Campinas, Brazil (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIS-01FOP
Record Dates: First submitted 2016-01-20; First posted 2016-02-02 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Anxiety; Pain
Keywords: nitrous oxide; conscious sedation; pain; anxiety
MeSH Terms: conditions — Anxiety Disorders; Pain | interventions — Nitrous Oxide; Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nitrous oxide (Experimental): Nitrous oxide sedation
  Interventions: Drug: Nitrous Oxide

INTERVENTIONS:
Drug: Nitrous Oxide — The N2O/O2 equipment was composed by two flow meters with an anti-hypoxia system valve, 70% N2O maximum disposal and 30 L/min O2 valve to immediate oxygen dispensation. Masks were individually selected, being 100% O2 (6 L/min) dispensed until respiratory rate stabilization. N2O was incremented at 10% each 2 minutes (70% max, if necessary) until some of the following signals were noticed: silence, relax/comfort report, decreased eyelid movements, decreased spontaneous body movements, warm sensation, tingling sensation or numbness at feet, hands or oral region, and slightly euphoric sensation.
  Other Names: Nitrous oxide / oxygen

SUMMARY:
BACKGROUND: The degree of consciousness during nitrous oxide use is still a matter of concern for both dentists and anesthesiologists. Investigators hypothesized that BIS levels do not vary according nitrous oxide concentration during minimum to moderate sedation in the dental treatment.

METHODS: One hundred patients undergoing dental procedures demanding local anesthesia (1.8 mL of 2% lidocaine with 1:100.000 epinephrine) were enrolled in this study. Initial pain and anxiety were measured by 11-point numerical and anxiety visual scales, respectively. Systolic/diastolic arterial blood pressure, SpO2, heart and respiratory rates, and psychomotor ability (Trieger test) were assessed before, during and after dental treatment. Sedation levels were evaluated by both BIS and sedation analogic scale at the same intervals. The duration of treatment along with nitrous oxide concentration and side effects were observed. Kruskal-Wallis, Friedman and Mann-Whitney tests were used (alpha=5%).

DETAILED DESCRIPTION:
One-hundred ASA I / II volunteers of both genders were selected in different dental speciality clinics (restorative dentistry, endodontics, implantology, and oral surgery) of Dental Institute of Pontifical Catholic University of Rio de Janeiro PUC-Rio).

After anamnesis and obtaining written informed consent, all volunteers were asked to fill an 11-point numerical scale in order to quantify the initial pain. The scale showed 0 as "no pain" and 10 as the "worst pain imaginable". In addition, volunteers were also asked to fill a facial image scale in order to determine the initial anxiety. This scale showed four levels: 0 corresponding to absolutely calm; 1 - slightly stressed; 2 - stressed; and 3 - extremely stressed.

The volunteers were positioned in the dental chair and instructed to fill a Trieger test (psychomotor evaluation) during the following periods: 1) before sedation; 2) during the sedation (10 minutes after respiratory stabilization with N2O/O2); and 3) 10 minutes after the end of sedation. The number of wrong connected points (precision) and the time required to fill all points were used to estimate psychomotor ability.

A pulse oxymeter was placed in the volunteers' thumb and an electronic sphygmomanometer was positioned in the forearm in order to evaluate oxygen saturation (SpO2), systolic and diastolic pressures, and hearth rate during the same moments of the Trieger test. Respiratory rate was evaluated at same moments, by direct observation of thoracic movements.

The electrodes of BIS monitor were placed and the values were obtained at same operatory periods previously described, despite the continuous BIS monitoring. After BIS-signal stabilization, the dental procedure and the sedation with N2O/O2 were explained to the volunteer. Two previously calibrated operators installed BIS electrodes, applied the Trieger test and sedated all subjects. A third operator performed the dental treatments.

Five minutes after reaching ideal sedation level, the anesthetic solution (1.8 mL of 2% lidocaine with 1:100.000 epinephrine) was injected. Right after the end of clinical procedure, 100% O2 were provided during 5 minutes and a new Trieger test was filled out. The volunteer was dismissed if this last Trieger test was compatible with the first one. At this moment, they were also asked about discomfort or complications. The duration and type of dental procedure were also registered.

The N2O/O2 equipment was composed by two flow meters with an anti-hypoxia system valve, 70% N2O maximum disposal and 30 L/min O2 valve to immediate oxygen dispensation. Masks were individually selected, being 100% O2 (6 L/min) dispensed until respiratory rate stabilization. N2O was incremented at 10% each 2 minutes (70% max, if necessary) until some of the following signals were noticed: silence, relax/comfort report, decreased eyelid movements, decreased spontaneous body movements, warm sensation, tingling sensation or numbness at feet, hands or oral region, and slightly euphoric sensation. The dental procedure started after 5 min from the ideal sedation achievement.

The sedation level was scored by using the five-points Observer's Assessment of Alertness/Sedation (OAA/S) scale, previously described elsewhere. In addition, BIS was used to monitoring brain cortical activity at 0.5 to 30 Hz frequency bandwidth, checking impedance before every reading. Impedance remained below 800 ohms. Zipprep-type electrodes were placed according to manufacturer instructions. Fp1-Fpz was monitored in channel 1, Fp2-Fpz in channel 2 and the ground reference was placed on the pre-auricular region. BIS and both BIS channel waves were recorded from successive 2 seconds periods 13 and updated at every 5 seconds. The automatic artifact detection and rejection system of the BIS monitor were used. Baseline levels were obtained before sedation.

Results were submitted to Kruskal-Wallis' (Dunn), Friedman's, Mann-Whitney's and Spearman's correlation tests. The significance level was set at 5%. The analysis was performed by using BioEstat 5.0.

ELIGIBILITY:
Inclusion Criteria:

* Any gender;
* Age from 18 to 60 years;
* Needing one or more specialized treatment, such as restorative dentistry, endodontics, implantology, or oral surgery.

Exclusion Criteria:

* Compulsive personality;
* Claustrophobia;
* Severe personal disorders;
* Chronic obstructive pulmonary diseases;
* Recent ear surgery history;
* Use of bleomycin during the last year;
* Use of CNS depressants;
* Use of analgesics or anti-inflammatory agents one week before the study;
* Former drug addicts;
* Pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2006-11; Primary Completion 2007-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
BIS value | two hours
  Relative values continuously registered by the BIS device

SECONDARY OUTCOMES:
Pain | two hours
  11-point numerical scale used to quantify the initial pain. The scale showed 0 as "no pain" and 10 as the "worst pain imaginable".
Anxiety | two hours
  Volunteers were asked to fill a facial image scale in order to determine the initial anxiety. This scale showed four levels: 0 corresponding to absolutely calm; 1 - slightly stressed; 2 - stressed; and 3 - extremely stressed.
Blood Pressure | two hours
  Measurement of blood pressure during two hours.
Heart rate | two hours
  Measurement of heart rate during two hours.
Respiratory Frequency (RF) | two hours
  Measurement of RF during two hours.
Trieger test | two hours
  Measurement of the lost points and time necessary for completion.

IPD SHARING:
Plan to Share IPD: No